CLINICAL TRIAL: NCT04404010
Title: Effectiveness of Immersive Virtual Reality Training Compared to Instructional Technical Surgical Video: A Randomized Controlled Trial
Brief Title: Virtual Reality vs Technical Video in Surgical Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: PrecisionOS Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20200008-01H
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Surgical Training
Keywords: Immersive Virtual Reality; Technical Training Video

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality (Active Comparator): Participants randomized to the immersive virtual reality (iVR) study arm, considered the "intervention group" will receive training on completion of a reverse shoulder arthroplasty using an iVR simulator (PrecisionOS Technology).
  Interventions: Other: Immersive Virtual Reality
- Surgical Video (Other): Participants randomized to the standard video study arm, considered the "control group" will receive training on completion of reverse shoulder arthroplasty using a technical surgical instructional video.
  Interventions: Other: Surgical Technical Instructional Video

INTERVENTIONS:
Other: Immersive Virtual Reality — Participants randomized to the iVR simulator utilizes a head-mounted display producing 3D visuals with haptic controllers for an immersive operating room experience. The module produced consists of the key steps in performing a reverse shoulder arthroplasty using virtual versions of the equipment used in the real procedure. Prior to initiation, participants will be provided with a safety and training demonstration on the use of the VR module by study personnel. Participants will be provided as much time as they require to watch the video, including repetition if desired, which they will be timed for completion.
  Arms: Immersive Virtual Reality
Other: Surgical Technical Instructional Video — Participants will be provided as much time as they require to watch the instructional video, including repetition if desired, which they will be timed for completion.
  Arms: Surgical Video

SUMMARY:
The use of instructional technical surgical videos is common in orthopaedic education. Many residents have used instructional technical surgical training videos prior to medical school, as well as during their residency program, and at instructional courses. The use of instructional technical surgical videos and multimedia is considered an adjunctive training method for orthopaedic residents to learn operative procedures.

Immersive virtual reality (iVR) is increasingly used in surgical education. Recently, iVR has shown transfer of skill training in orthopaedics. The continued study of the effectiveness of iVR training in orthopaedic education could benefit new competency based orthopaedics residency programs.

The purpose of this study is to compare the effectiveness of instructional technical surgical video training to immersive iVR training for teaching technical skills of reverse total shoulder arthroplasty. Our hypothesis was that iVR improved learning effectiveness compared to standard technical surgical video. Secondary objectives include validating a virtual reality ratings scale through correlation to real-world performance.

We proposed a randomized, blinded intervention-control trial directly comparing immersive iVR versus technical surgical instructional video training in the teaching of reverse shoulder arthroplasty in senior residents, learning at the 2020 annual Canadian Shoulder and Elbow Society meeting.

DETAILED DESCRIPTION:
The use of instructional technical surgical videos is common in orthopaedic education. Many residents have used instructional technical surgical training videos prior to medical school, as well as during their residency program, and at instructional courses. The use of instructional technical surgical videos and multimedia is considered an adjunctive training method for orthopaedic residents to learn operative procedures.

Immersive virtual reality (iVR) is increasingly used in surgical education. Recently, iVR has shown transfer of skill training in orthopaedics. The continued study of the effectiveness of iVR training in orthopaedic education could benefit new competency based orthopaedics residency programs.

The purpose of this study is to compare the effectiveness of instructional technical surgical video training to immersive iVR training for teaching technical skills of reverse total shoulder arthroplasty. Our hypothesis was that iVR improved learning effectiveness compared to standard technical surgical video. Secondary objectives include validating a virtual reality ratings scale through correlation to real-world performance, and to determine efficiency of learning in both groups.

Currently, technical surgical instructional videos are pervasive in orthopaedic teaching education. Immersive VR, another form of teaching, is increasingly being used in surgical education. The production of an immersive VR suite with tactile and user metric feedback may be an advance over current bench top simulator technology, allowing for greater immersion and interaction, leading to better understanding of surgical planning and implementation. The development of this technology could provide trainees with immersive levels of training not previously seen, with improved learning of technical skills over media such as manufacturer technical documents. The effectiveness of training and efficiency of training of the novel immersive VR training systems need to be evaluated as they are increasingly incorporated into competency based, contemporary residency education.

We proposed a randomized, blinded intervention-control trial directly comparing immersive iVR versus technical surgical instructional video training in the teaching of reverse shoulder arthroplasty in senior (fourth and fifth year) residents, learning at the 2020 annual Canadian Shoulder and Elbow Society meeting.

ELIGIBILITY:
Inclusion Criteria:

* Senior residents (4th and 5th year residents) attending 2020 CSES course

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Pollock, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The University of Ottawa Skills and Simulation Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lohre R, Bois AJ, Pollock JW, Lapner P, McIlquham K, Athwal GS, Goel DP. Effectiveness of Immersive Virtual Reality on Orthopedic Surgical Skills and Knowledge Acquisition Among Senior Surgical Residents: A Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2031217. doi: 10.1001/jamanetworkopen.2020.31217. PMID 33369660

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was mistakenly consented (error in screening - participant was not a PGY4 or 5) and randomized to immersive virtual reality arm as part of study. After randomization, but prior to study testing we realized the participant was not eligible, therefore they were excluded prior to any further study procedures commenced.
  1 additional participant was mistakenly consented (error in screening - participant was not a PGY4 or 5), therefore excluded PRIOR to randomization.
Period: Overall Study
Arm/Group | Immersive Virtual Reality | Surgical Video
Started | 10 (1 participant was mistakenly consented, enrolled and randomized as part of study. After randomization, but prior to study testing we realized the participant was not eligible (they were not a PGY4 or 5), therefore they were excluded prior to any further study procedures commenced. Therefore, only 9 participants completed all study procedures/were followed for purposes of study.) | 9
Completed | 9 | 9
Not Completed | 1 | 0
Not completed — Mistakenly enrolled, withdrawn after randomization (did not meet eligibility criteria) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immersive Virtual Reality | Surgical Video | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Structured Assessment of Technical Skills (OSATS)
Description: The Objective Structured Assessment of Technical Skills (OSATS) outcome measure is a validated assessment tool used for grading overall technical ability during surgery. This checklist contains 27 items, in which an assessor will mark off whether the task was completed successfully or not. For each item done correctly, it is worth 1 point. For each item done incorrectly, no point is awarded. All points are totalled for a maximum possible score of 27 points (minimum score of 0 and maximum score of 27). A higher score indicates a better outcome.
Time Frame: During surgery up until immediately after surgery.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immersive Virtual Reality | Surgical Video
Number analyzed (Participants) | 9 | 9
score on a scale | 15.9 [14.3 to 17.5] | 9.4 [7.4 to 11.5]

2. Secondary Outcome: Global Ratings Scale (GRS)
Description: The Global Ratings Scale (GRS) is a validated assessment tool used for grading operative performance. The GRS contains 7 categories: respect for tissue, time and motion, instrument handling, knowledge of instruments, flow of operation, use of assistants, and knowledge of specific procedure. Each category is graded using a 5-point Likert type scale, a higher number indicates a better outcome, with a maximum of 5 points per category. Each categorical score is totalled for a maximum overall score of 35 points (minimum score of 0 and maximum score of 35). A higher score indicates a better outcome.
Time Frame: During surgery up until immediately after surgery.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immersive Virtual Reality | Surgical Video
Number analyzed (Participants) | 9 | 9
Score on a scale | 22.8 (8.2) | 22.4 (9.0)

3. Secondary Outcome: Transfer of Training (ToT)
Description: Transfer of Training (ToT) outcome informs how much skill is gained in the iVR group compared to the control performance. This is measured using an equation. ToT equals the average time to complete surgical procedure (for those in instructional video group) minus the average time to complete the surgical procedure (for those in the iVR training group), divided by the average time to complete surgical procedure (for those in instructional video group). The outcome is presented as a cumulative ratio, and a numerical value is provided. A higher number indicates a better outcome. For the purpose of this project, there is not a spread of data for a single instance of training as we did not complete multiple repetitions, otherwise we would have incremental values for each.
Time Frame: immediately after surgery.
Population: The ToT is calculated as a cumulative ratio. There isn't a spread of data for a single instance of training, however, if we had done more repetitions then we would have incremental values for each. Therefore, the single numerical value of ToT is 0.594 or 59.4%. Answer is based off of the following calculation: (Time (surgical video) - Time (immersive virtual reality) divided by the Time (surgical video)) multiplied by 100%.
Measure: Mean (Full Range); unit: Percentage
Groups:
- Transfer of Training Ratio: A comparison of skill achievement compared to control performance. This informs how much skill is gained by training.
Arm/Group | Transfer of Training Ratio
Number analyzed (Participants) | 18
Percentage | 59.4 [0 to 100]

4. Secondary Outcome: Transfer Effectiveness Ratio (TER)
Description: Transfer Effectiveness Ratio (TER) outcomes informs on the skill comparison relative to the control, on real world training reduction times. TER equals the average time to complete surgical procedure (for those in instructional video group) minus the average time to complete the surgical procedure (for those in the iVR training group), divided by the average time to complete the iVR training. The outcome is presented as a cumulative ratio, and a numerical value is provided. A higher number, indicates a better outcome. For the purpose of this project, there is not a spread of data for a single instance of training as we did not complete multiple repetitions, otherwise we would have incremental values for each.
Time Frame: Immediately before surgery up immediately after surgery.
Population: The TER is calculated as a cumulative ratio. There isn't a spread of data for a single instance of training, however, if we had done more repetitions then we would have incremental values for each. Therefore, the single numerical value of TER is 0.79. Answer is based off of the following calculation: (Time (surgical video) - Time (immersive virtual reality) divided by Time (simulated immersive virtual reality)).
Measure: Mean (Full Range); unit: Ratio Value
Groups:
- Transfer Effectiveness Ratio: Skill comparison relative to control, incorporating improvements in task time. This informs real world training reduction times.
Arm/Group | Transfer Effectiveness Ratio
Number analyzed (Participants) | 18
Ratio Value | 0.79 [0 to 1.0]

ADVERSE EVENTS:
Time Frame: 1 day (duration of each participant's involvement in study)
Description: There are no serious risks associated with this study. The purpose of this study was to compare training methods to determine which one is most effective among orthopaedic surgical residents. There was a possibility for those in the virtual reality group to experience dizziness or nausea, however is considered mild and rare. Trained personnel were available to assist throughout the duration of training as well.
Arm/Group | Immersive Virtual Reality | Surgical Video
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT04404010/Prot_SAP_000.pdf